CLINICAL TRIAL: NCT04318093
Title: A Randomized, Double-Blinded, Placebo-Controlled, Study to Evaluate the Safety and Tolerability of BMS-986259 in Stabilized Patients Hospitalized for Acute Decompensated Heart Failure
Brief Title: Study of the Safety of BMS-986259 in Participants With Post-Acute Decompensated Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CV019-010; 2019-004186-40 (EudraCT Number)
Record Dates: First submitted 2020-03-20; First posted 2020-03-23 (Actual); Results first posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Acute Decompensated Heart Failure
Keywords: Heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BMS-986259 (Experimental)
  Interventions: Drug: BMS-986259
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BMS-986259 — Specified dose on specified days
  Arms: BMS-986259
Other: Placebo — Specified dose on specified days
  Arms: Placebo

SUMMARY:
The purpose of the study is to assess the safety of BMS-986259 in stable participants hospitalized for acute decompensated heart failure.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Participants currently hospitalized for acute decompensated heart failure (ADHF)
* Participants must be hemodynamically stable, as assessed by the investigator
* Men must agree to follow specific methods of contraception, if applicable, while participating in the trial
* Women participants must have documented proof that they are not of childbearing potential

Exclusion Criteria:

* Acute cardiovascular condition other than heart failure (HF) decompensation
* Cardiogenic shock at presentation to emergency room (ER) or at any time before randomization
* Recipient of ventricular assist devices or use of any cardiac extracorporeal devices, within 12 weeks of study randomization
* Participants with contraindications to vasodilator therapy such as restrictive or obstructive cardiomyopathy, severe mitral or aortic stenosis

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2021-07-19 (Actual); Study Completion 2021-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (18):
- Argentina (6):
  - Local Institution - 0009, Ciudad de Buenos Aires, Buenos Aires
  - Local Institution - 0007, Alberdi, Córdoba Province
  - Local Institution - 0028, Córdoba, Córdoba Province
  - Local Institution - 0010, Córdoba, Córdoba Province
  - Local Institution, Buenos Aires, Distrito Federal
  - Local Institution - 0025, Córdoba
- Czechia (2):
  - Local Institution - 0020, Prague
  - Nemocnice Slany-Interna - kardiologicka ambulance, Slaný
- Greece (2):
  - Local Institution - 0011, Athens
  - Local Institution - 0022, Athens
- Israel (3):
  - Local Institution - 0014, Tel Aviv, Tell Abīb
  - Local Institution, Jerusalem
  - Local Institution, Petah Tikva
- Poland (3):
  - Local Institution - 0034, Bialystok
  - Local Institution - 0030, Wrocaw
  - Local Institution - 0027, Wroclaw
- United Kingdom (2):
  - Local Institution, Edinburgh
  - Local Institution, Swindon

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 25 participants were randomized and treated.
Groups:
- Placebo: Placebo matching BMS-986259
- BMS-986259 3 mg: BMS-986259 administered subcutaneously QD for 14 days
Period: Overall Study
Arm/Group | Placebo | BMS-986259 3 mg
Started | 13 | 12
Completed | 10 | 9
Not Completed | 3 | 3
Not completed — Adverse Event | 2 | 2
Not completed — Participant withdrew consent | 1 | 0
Not completed — Other reasons | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BMS-986259 3 mg | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 6 | 10
  >=65 years | 9 | 6 | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.1 (12.18) | 63.1 (15.65) | 64.1 (13.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 9 | 9 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 12 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Clinically Relevant Hypotension
Description: Clinically Relevant Hypotension is defined as occurrence of any of the following:
  * Supine Systolic Blood Pressure (SBP) <85 mmHg (confirmed by repeat measurement within 30 minutes), regardless of symptoms of hypotension
  * Supine SBP <90 mmHg (confirmed by repeat measurement within 30 minutes) AND symptoms of hypotension (eg, dizziness, lightheadedness, etc).
Time Frame: From first dose to 30 days following first dose
Population: All treated participants
Measure: Number; unit: Percent of participants
Arm/Group | Placebo | BMS-986259 3 mg
Number analyzed (Participants) | 13 | 12
Percent of participants | 15.4 | 16.7

2. Secondary Outcome: Maximum Observed Serum Concentration (Cmax)
Time Frame: Day 1 and Day 5 of study treatment
Population: All participants receiving study drug with available measurements
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | BMS-986259 3 mg
Number analyzed (Participants) | 12
ng/mL
  Day 1 | 105 (49)
  Day 5: number analyzed (Participants) | 9
  Day 5 | 268 (31)

3. Secondary Outcome: Time of Maximum Observed Serum Concentration (Tmax)
Time Frame: Day 1 and Day 5 of study treatment
Population: All participants receiving study drug with available measurements
Measure: Median (Full Range); unit: Hours
Arm/Group | BMS-986259 3 mg
Number analyzed (Participants) | 12
Hours
  Day 1 | 11.0 [7.00 to 23.3]
  Day 5: number analyzed (Participants) | 9
  Day 5 | 7.97 [5.00 to 24.0]

4. Secondary Outcome: Area Under the Concentration-Time Curve Within a Dosing Interval (AUC(TAU))
Time Frame: Day 1 and Day 5 of study treatment
Population: All participants receiving study drug with available measurements
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | BMS-986259 3 mg
Number analyzed (Participants) | 9
h*ng/mL
  Day 1 | 1778 (40)
  Day 5: number analyzed (Participants) | 7
  Day 5 | 5156 (36)

5. Secondary Outcome: Trough Concentration (Ctrough)
Time Frame: Day 2 through Day 14 of study treatment (with the exception of Day 11, for which data is not available)
Population: All participants receiving study drug with available measurements
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | BMS-986259 3 mg
Number analyzed (Participants) | 11
ng/mL
  Day 2: number analyzed (Participants) | 9
  Day 2 | 79.9 (36.0)
  Day 3 | 145 (32.3)
  Day 4: number analyzed (Participants) | 7
  Day 4 | 181 (28.9)
  Day 5: number analyzed (Participants) | 10
  Day 5 | 185 (32.4)
  Day 6: number analyzed (Participants) | 7
  Day 6 | 210 (27.3)
  Day 7: number analyzed (Participants) | 6
  Day 7 | 260 (41.3)
  Day 8: number analyzed (Participants) | 8
  Day 8 | 226 (69.4)
  Day 9: number analyzed (Participants) | 5
  Day 9 | 252 (48.1)
  Day 10: number analyzed (Participants) | 5
  Day 10 | 259 (49.7)
  Day 12: number analyzed (Participants) | 4
  Day 12 | 229 (22.9)
  Day 13: number analyzed (Participants) | 5
  Day 13 | 248 (50.5)
  Day 14: number analyzed (Participants) | 3
  Day 14 | 246 (7.53)

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from first dose to study completion date (up to approximately 8 months). SAEs and NSAEs were assessed from first dose to 30 days following first dose.
Groups:
- BMS986259 3 mg: BMS-986259 administered subcutaneously QD for 14 days
Arm/Group | Placebo | BMS986259 3 mg
All-Cause Mortality (participants affected / at risk) | 2/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 5/13 | 2/12
Other Adverse Events (participants affected / at risk) | 3/13 | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=13) | BMS986259 3 mg (N=12)
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
COVID-19 (Infections and infestations) | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=13) | BMS986259 3 mg (N=12)
Haemoconcentration (Blood and lymphatic system disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Genital haemorrhage (Reproductive system and breast disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-28): https://cdn.clinicaltrials.gov/large-docs/93/NCT04318093/Prot_SAP_000.pdf